CLINICAL TRIAL: NCT01040806
Title: Peer Coaching for Low-Income Patients With Diabetes in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: American Academy of Family Physicians (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H40013-34104-01
Record Dates: First submitted 2009-12-28; First posted 2009-12-30 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Type 2
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health coaching (Experimental): Patients with poorly controlled diabetes will receive counseling from a peer health coach -- a patient with diabetes trained in health coaching
  Interventions: Behavioral: Health coaching
- Usual care (Active Comparator): Patients will receive usual care
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Usual care — Patients will receive their usual medical care
  Arms: Usual care
Behavioral: Health coaching — Peer health coaches will counsel patients with diabetes
  Other Names: Peer coaching; Peer coach; Peer support
  Arms: Health coaching

SUMMARY:
Patients with diabetes who are counseled by a peer coach (another patient with diabetes) will have improved glycemic control compared with usual care patients.

DETAILED DESCRIPTION:
Peer coaches have controlled diabetes, patient study subjects have poorly controlled diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes with most recent HbA1c 8 or above in past 6 months.

Exclusion Criteria:

* Dementia,
* Life expectancy less than 6 months,
* Inability to speak English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2009-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
HbA1c level | 6 months

SECONDARY OUTCOMES:
LDL cholesterol level | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bodenheimer, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Background] Ghorob A, Vivas MM, De Vore D, Ngo V, Bodenheimer T, Chen E, Thom DH. The effectiveness of peer health coaching in improving glycemic control among low-income patients with diabetes: protocol for a randomized controlled trial. BMC Public Health. 2011 Apr 1;11:208. doi: 10.1186/1471-2458-11-208. PMID 21457567
- [Derived] Thom DH, Ghorob A, Hessler D, De Vore D, Chen E, Bodenheimer TA. Impact of peer health coaching on glycemic control in low-income patients with diabetes: a randomized controlled trial. Ann Fam Med. 2013 Mar-Apr;11(2):137-44. doi: 10.1370/afm.1443. PMID 23508600